CLINICAL TRIAL: NCT06820593
Title: Technology-Enhanced Asthma Care in Children at Clinic and Home (TEACCCH) Study (Aim 2): A Feasibility Randomized Controlled Trial
Brief Title: Technology-Enhanced Asthma Care in Children at Clinic and Home Study
Acronym: TEACCCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kristin Kan, Assistant Professor, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-6333; K23HL157615 (NIH)
Record Dates: First submitted 2025-01-24; First posted 2025-02-11 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Asthma in Children; Chronic Diseases in Children
Keywords: Digital Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Asthma Intervention (Experimental): The intervention group will receive digital tools (mHealth app and sensors) and remote patient monitoring (RPM) assisted by an asthma coordinator, that supports an enhanced standard of care for their child's asthma. The mHealth intervention includes inhaler sensors on their rescue (SABA) and ICS inhaler and a mHealth app on the parent's smartphone. The asthma coordinator, as part of the implementation plan, will respond to information from the mHealth app and contact the participants about their adherence and asthma symptom control, following an algorithm aligned with NAEPP guidelines.
  Interventions: Behavioral: Digital Asthma Intervention
- Comparison (Active Comparator): The comparison group will also receive enhanced standard of asthma care. A research "control" version of the mHealth app will be downloaded to smartphones to allow for data collection from inhaler sensors, but the mHealth app will only silently transmit data to the web portal and not provide any app interaction or feedback to participants.
  Interventions: Behavioral: Comparison Group

INTERVENTIONS:
Behavioral: Digital Asthma Intervention — The intervention consists of two main components-the mHealth app and sensors that is part of the Adherium's Hailie® Solution-and the remote patient monitoring (RPM), conducted in this intervention by an asthma coordinator.
  Arms: Digital Asthma Intervention
Behavioral: Comparison Group — Participants in the comparison group will receive the sensors for their ICS inhalers and a limited version of the app that only collects the sensor information by Bluetooth, without app features, and sends the information to the Hailie web portal. This passive adherence data collection will allow for comparison of the two groups' adherence rates without the mHealth app self-management support or RPM.
  Arms: Comparison

SUMMARY:
A randomized controlled trial with parent-child pairs of children with persistent or uncontrolled asthma. An intervention group (n=40 parent-child pairs) will receive the mobile health (mHealth) app and digital sensors with enhanced support from a population health manager role, hereinafter referred to as an asthma coordinator, to provide remote patient monitoring (RPM). A comparison group (n=40 parent-child pairs) will receive the mHealth app and sensors without RPM support to silently collect inhaler use information without mHealth app features. The focus of this project is to evaluate the feasibility and acceptability of delivering a digital intervention for pediatric asthma with RPM in the outpatient setting.

ELIGIBILITY:
Inclusion into the study will not depend on sex, ethnicity, or race. We will monitor enrollment to ensure a diversity of sex and race/ethnicity are represented.

PARENT-CHILD PAIR INCLUSION CRITERIA

1. Caregivers must be at least 18 years old (defined as parent or legal guardian)
2. The child (patient) has a diagnosis of asthma associated with a clinic visit in the electronic health record
3. The child is between the ages of 4-17 years old at the time of recruitment

   1. The study is interested in the self-management of asthma by caregivers, whom are still primarily responsible for their child's chronic disease management.
   2. Children younger than 4 years old will not be included in this study as the diagnosis of asthma is typically difficult to confirm in younger ages.
4. The child is prescribed inhaled corticosteroid or corticosteroid/long-acting beta agonist combination for daily use. The patient can have an inhaled corticosteroid/long-acting beta agonist for both daily preventive and rescue use, as in Single Maintenance and Reliever Therapy (SMART).
5. Persistent or un controlled asthma based on NHLBI guidelines40; Any 1 of the following:

   1. In past month, >2 days per week with asthma symptoms
   2. >2 days per week with rescue medication use
   3. >2 days per month with nighttime awakenings (for children who are not taking a controller asthma medication) OR >2 days per month with nighttime awakenings (for children who are currently taking a controller asthma medication)
   4. >2 asthma episodes during the past year that required systemic corticosteroids
6. The child is a patient in Primary Care Uptown, Primary Care Deming, Allergy, or Pulmonary Clinics at LCH

PARENT-CHILD PAIR EXCLUSION CRITERIA

1. The caregiver has a smartphone that is not compatible with the Hailie® app.
2. The patient is prescribed a controller (preventive) or rescue inhaler medication to which the Hailie electronic sensor cannot affix.
3. The caregiver is unable to speak and understand English.

   a. With this trial, the intent is to first establish feasibility and broaden to different languages in future.
4. The child has clinically significant, comorbid diagnoses, such as cystic fibrosis, cyanotic heart disease, or bronchopulmonary dysplasia, that could interact with their assessment of asthma-related measures.
5. The family has active Department of Child and Family Services (DCFS) involvement
6. The participant is enrolled in another asthma intervention study at the time of enrollment to this study.
7. Child or sibling living in the same home was previously enrolled in this study.
8. Consent is not obtained from the parent/guardian.
9. Parent/guardian does not pass the test of understanding at study enrollment.

HEALTH CARE PROVIDER INCLUSION CRITERIA (IMPLEMENTATION OUTCOMES)

1. Participant is an employee of LCH system
2. Works at or supports the operations of Primary Care Uptown, Primary Care Deming, Allergy, or Pulmonary Clinics at LCH
3. Able to provide informed consent

HEALTH CARE PROVIDER EXCLUSION CRITERIA (IMPLEMENTATION OUTCOMES)

1. Participant departs LCH and is no longer an active employee at the time of assessment

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Study Feasibility | Baseline, 12 months
  Measured as the number and percentage of participants who complete the 12-month visit, between intervention and comparison group.

SECONDARY OUTCOMES:
Intervention Feasibility | 12 months
  Measured as the number and percentage of participants who synced their ICS sensor >80% of enrolled days in the trial, comparing intervention and comparison groups.
Asthma Symptom Control | Baseline, 1, 3, 6, 9, and 12 months.
  Investigators will use the validated childhood Asthma Control Test (c-ACT) for assessing asthma symptom control, or Asthma Control Test (ACT) if the child becomes 12 years old during the study.
Inhaled Corticosteroid Adherence | Continuously through the 12 months
  Investigators will compare overall raw ICS adherence rates between intervention and comparison groups using two-sample tests for proportions of mean daily proportion of taken doses over prescribed doses of ICS by study month, measured by digital sensors on the ICS. Participants' data will be included if they had at least 1 ICS inhaler actuation during the trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States